CLINICAL TRIAL: NCT02013232
Title: Adjunctive Aripiprazole in the Treatment of Risperidone-Induced Hyperprolactinemia: A Randomized, Double-Blind, Placebo-Controlled, Dose-Response Study
Brief Title: Adjunctive Aripiprazole in the Treatment of Risperidone-Induced Hyperprolactinemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Jingxu Chen, associate professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI201206
Record Dates: First submitted 2013-12-02; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia
Keywords: Risperidone;; Aripiprazole;; Hyperprolactinemia;; dose effects
MeSH Terms: conditions — Schizophrenia; Hyperprolactinemia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo (Placebo Comparator): risperidone plus placebo
- aripiprazole 5mg (Experimental): risperidone treatment plus aripiprazole 5mg/day
  Interventions: Drug: Aripiprazole
- aripiprazole 10mg (Experimental): risperidone plus aripiprazole 10mg/day
  Interventions: Drug: Aripiprazole
- aripiprazole 20mg (Experimental): risperidone plus aripiprazole 20mg/day
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole
  Arms: aripiprazole 10mg; aripiprazole 20mg; aripiprazole 5mg

SUMMARY:
Hyperprolactinemia is a frequent consequence of treatment with typical antipsychotic agents and atypical antipsychotics such as risperidone. Recent studies have suggested that aripiprazole, a partial dopamine agonist, reduces the prolactin response to antipsychotics. Thus, we conducted this study to evaluate the dose effects of adjunctive treatment with aripiprazole on hyperprolactinemia in stable schizophrenic patients maintained with risperidone.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-45 years of and fulfilled Diagnostic and Statistical Manual of Mental Disorders(DSM-IV )criteria (American Psychiatric Association, 1994) for schizophrenia;
2. having a stable psychiatric condition, defined as taking the same dosage of risperidone for at least 6 weeks;
3. being treated with risperidone monotherapy; and presence of hyperprolactinemia associated with risperidone.

Exclusion Criteria:

1. any other major psychiatric disorder;
2. significant concurrent medical illnesses, organic brain disorder, history of substance and alcohol abuse, and mental retardation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Prolactin level | baseline, 2 weeks, 4 weeks, 8 weeks
  Change from baseline in the levels of prolactin

SECONDARY OUTCOMES:
PANSS (positive and negative syndrome scale) score | Baseline, 8 weeks
  Change from baseline in PANSS score

OTHER OUTCOMES:
extrapyramidal symptoms | baseline, 4 weeks, 8 weeks
  assess the extrapyramidal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality, China